CLINICAL TRIAL: NCT05519176
Title: A Study of Risk Factors for Venous Ulceration in Patients With Varicose Veins of Lower Extremities: A Case-control Study.
Brief Title: A Study of Risk Factors for Venous Ulceration in Patients With Varicose Veins of Lower Extremities.
Status: Completed | Type: Observational
Sponsor: Yibing Wang (Other)
Responsible Party: Sponsor-Investigator, Yibing Wang, professor, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: YXLL-KY-2022(053)
Record Dates: First submitted 2022-08-26; First posted 2022-08-29 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Venous Ulceration
Keywords: Varicose Veins; Varicose Ulcer; Leg Ulcer; Case-Control Study
MeSH Terms: conditions — Varicose Ulcer; Varicose Veins; Leg Ulcer

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Varicose veins of lower extremities inpatients with venous ulceration from The First Affiliated Hospital of Shandong First Medical University & Shandong Provincial Qianfoshan Hospital.
- Controls: Varicose veins of lower extremities inpatients without venous ulceration from The First Affiliated Hospital of Shandong First Medical University & Shandong Provincial Qianfoshan Hospital.

SUMMARY:
Varicose veins of lower extremities can lead to adverse consequences such as ulceration and hemorrhage, which seriously endangering the physical and mental health and quality of life for patients.

The aim of this study is to explore the potential risk factors of venous ulceration in patients with varicose veins of lower extremities based on a case-control study, and to provide a reference for personalized treatment.

DETAILED DESCRIPTION:
Varicose veins of lower extremities are common chronic diseases. The main clinical manifestations are lower extremity weakness, heaviness, burning sensation, itching, swelling or pain, and severe cases are often accompanied by complications such as changes in skin color, ulceration and hemorrhage. Venous ulceration is one of the main complications of lower extremity varicose veins, accounting for more than 75% of all lower extremity ulcers. Venous ulceration are difficult to heal and prone to recurrence. Studies have shown that the recurrence rate of venous ulceration is as high as 67%. The refractory and high recurrence rate of venous ulceration not only have a serious impact on the quality of patients' life, but also bring a heavy economic burden on society.

Venous ulceration in varicose veins of lower extremities patients may linked to different causes, including past medical history, comorbidity, inflammatory response, etc. The purpose of this study is to collect demographic characteristics, lifestyle characteristics, laboratory indicators, past history, comorbidity and other information by using the data set of patients with varicose veins of lower extremities based on the Shandong Provincial Qianfoshan Hospital Healthcare Big Data Platform. To explore the potential risk factors of venous ulceration in patients with varicose veins of lower extremities through case-control study.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of varicose veins of the lower extremities
2. Hospitalized patients
3. 18 years old or older

Exclusion Criteria:

1. Patients with any other conditions that could also lead to venous ulceration including peripheral artery disease, diabetes, and pressure ulcers
2. Patients with heart, liver and kidney failure
3. Patients with malignant tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cases and controls are inpatients with varicose veins of lower extremities in The First Affiliated Hospital of Shandong First Medical University & Shandong Provincial Qianfoshan Hospital between January 1, 2016 and December 31, 2020.
Sampling Method: Non-Probability Sample
Enrollment: 1234 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Odds ratios of risk factors for venous ulceration | 2016-2020
  Age, gender, diastolic blood pressure, systolic blood pressure, routine blood indexes, coagulation indexes, duration of varicose veins of lower extremities, height, weight, smoking and drinking, comorbidity, family history of venous diseases, usage in anticoagulants and antihypertensives are all the possible risk factors of venous ulceration.

CONTACTS AND LOCATIONS:
Overall Officials: Wang Yibing, Doctor, Principal Investigator — The First Affiliated Hospital of Shandong First Medical University & Shandong Provincial Qianfoshan Hospital
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University & Shandong Provincial Qianfoshan Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided